CLINICAL TRIAL: NCT03927508
Title: First - In - Man Study to Assess the Safety and Feasibility of The Bashir™ Endovascular Catheter for the Treatment of Acute Pulmonary Embolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thrombolex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THRO-CLIN-2018-01
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Pulse Spray and Infusion of r-tPA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- BEC Treatment (Experimental): The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery.
  Interventions: Drug: r-tPA; Device: The Bashir™ Endovascular Catheter

INTERVENTIONS:
Drug: r-tPA — Pulse spray and infusion
Device: The Bashir™ Endovascular Catheter — The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature.

SUMMARY:
The Bashir™ Endovascular Catheter is a device intended for the localized infusion of therapeutic agents into the pulmonary artery and peripheral vasculature.

DETAILED DESCRIPTION:
The Bashir™ Endovascular Catheter has been designed to administer therapeutic agents in the peripheral vasculature. Because of the unique design of the catheter, with its six expandable infusion limbs, the Bashir™ Endovascular Catheter has the ability to: 1. Create a much larger central channel for blood flow, thereby utilizing the body's own endogenous fibrinolytic agents to lyse the clot, and 2. Greatly enhance the radial dispersion of a catheter-administered thrombolytic agent throughout the thrombus. Expansion of the multiple arms of the basket in the infusion catheter causes fissuring of the clot. The net result is that a greater surface area of clot is exposed to both endogenous and exogenously administered lytic agents, thereby promoting clot dissolution.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Willing and able to provide informed consent;
2. 18 years of age and less than 75 years of age;
3. PE symptom duration ≤ 14 days;
4. Filling defect in at least one main or lobar pulmonary artery as determined by contrast enhanced chest CT;
5. RV/LV end diastolic diameter ratio ≥ 0.9 by CTA as determined by the investigative site;
6. Willing and able to comply with all study procedures and follow-up.

Exclusion Criteria:

1. Cerebrovascular Accident (CVA) or transient ischemic attack (TIA) within one (1) year;
2. Head trauma, or other active intracranial, or intraspinal disease within one (1) year;
3. Recent (within one month) or active bleeding from a major organ;
4. Intracranial condition(s) that may increase the risk of bleeding (e.g., neoplasms, arteriovenous malformations, or aneurysms);
5. Patients with bleeding diathesis;
6. Hematocrit < 30%;
7. Platelets < 100,000/μL;
8. INR > 1.5;
9. aPTT > 50 seconds in the absence of anticoagulants;
10. Major surgery within fourteen (14) days;
11. Serum creatinine > 2 mg/dL;
12. Clinician deems high-risk for catastrophic bleeding;
13. History of heparin-induced thrombocytopenia (HIT);
14. Pregnancy;
15. Systolic blood pressure < 90 mmHg for > 15 minutes;
16. Any vasopressor support;
17. Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR);
18. Evidence of irreversible neurological compromise;
19. Life expectancy < one (1) year;
20. Use of thrombolytics or glycoprotein IIb/IIIa antagonists within 3 days prior to inclusion in the study;
21. Use of non-vitamin K oral anti-coagulants (NOACs), such as Rivaroxaban, Apixaban, Dabigatran, Edoxaban within 48 hours prior to inclusion in the study;
22. Use of enoxaparin sodium injection (Lovenox®) within 12 hours of procedure start time;
23. Profound bradycardia requiring a temporary pacemaker and/or inotropic support;
24. Previous enrollment in this study;
25. Morbidly obese (BMI >45 kg/m2) patient who by the judgement of the investigator is high risk for bleeding;
26. Absolute contraindication to anticoagulation;
27. Uncontrolled hypertension;
28. Currently participating in another study;
29. In the opinion of the investigator, the subject is not a suitable candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Advent Health Orlando, Orlando, Florida
  - St Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - Columbia University Medical Center - Presbyterian - New York, New York, New York
  - University Pittsburg Medical Center - Hamot, Erie, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sista AK, Bhatheja R, Rali P, Natarajan K, Green P, Piazza G, Comerota AJ, Parikh SA, Lakhter V, Bashir R, Rosenfield K. First-in-Human Study to Assess the Safety and Feasibility of the Bashir Endovascular Catheter for the Treatment of Acute Intermediate-Risk Pulmonary Embolism. Circ Cardiovasc Interv. 2021 Jan;14(1):e009611. doi: 10.1161/CIRCINTERVENTIONS.120.009611. Epub 2020 Dec 24. PMID 33356383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place over a period of four (4) months, July 19, 2019 - November 16, 2019. The date the study is was open for recruitment started March 14, 2019. Study was FDA approved for up to five (5) sites. Nine (9) subjects were enrolled and are included in this report through 30-day follow-up.
Period: Overall Study
Arm/Group | BEC Treatment
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BEC Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.67 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Major Bleeding Events
Description: Major Bleeding as defined by International Society of Thrombosis and Hemostasis (ISTH), within 72 hours of initiation of r-tPA administration. Bleeding criteria are as follows: Major Bleeding in Non-Surgical Patients
  1. Fatal bleeding; and/or
  2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome; and/or
  3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more or leading to transfusion of two or more units of whole blood or red cells.
Time Frame: Within 72 hours of initiation of r-tPA administration.
Measure: Count of Participants; unit: Participants
Arm/Group | BEC Treatment
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: From treatment through 30 days
Arm/Group | BEC Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEC Treatment (N=9)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEC Treatment (N=9)
Pain (General disorders) | 2 (2)
Tenderness (General disorders) | 2 (2)
Injection site pain (General disorders) | 1 (1)
occult blood (Investigations) | 1 (1)
tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Hypoaesthia (Nervous system disorders) | 1 (1)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Odema peripheral (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT03927508/Prot_SAP_000.pdf